CLINICAL TRIAL: NCT00814541
Title: Phase II Study to Assess the Safety, Efficacy, and Tolerability of Combination Therapy With Velcade (Bortezomib), Doxorubicin, and Dexamethasone (PAD) as Therapy for Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: PAD. ICORG 05-01, V11
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-01 ICORG; ICORG-05-01; 2005-000395-41; EU-20893; NCT00567138 (obsolete NCT alias)
Record Dates: First submitted 2008-12-24; First posted 2008-12-25 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-01

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: refractory multiple myeloma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Bortezomib; Doxorubicin; Dexamethasone

ARMS (3):
- 1 (Experimental): Relapsed patients, previously treated with VAD or VAD like regimen (VAMP, C-VAMP and Z-Dex are examples of VAD like therapy) and who have had autologous transplants at least 1 year previously.Patients may proceed directly to PAD therapy or have had a maximum of one other line of therapy before PAD.
  Interventions: Drug: Bortezomib; Drug: Doxorubicin; Drug: Dexamethasone
- 2 (Experimental): Relapsed patients, previously treated with VAD or VAD-like regimen who have not had autologous transplantation and achieved at least PR (Appendix A). Patients may proceed directly to PAD therapy or have had a maximum of two other lines of therapy before PAD.
  Interventions: Drug: Bortezomib; Drug: Doxorubicin; Drug: Dexamethasone
- 3 (Experimental): Patients refractory (MR, NC or PD) to VAD or VAD-like therapy. Patients should proceed directly to PAD therapy. Patients with NC or PD may proceed to PAD after a minimum of two cycles of VAD or VAD-like therapy or a minimum of 4 cycles, if MR.
  Interventions: Drug: Bortezomib; Drug: Doxorubicin; Drug: Dexamethasone

INTERVENTIONS:
Drug: Bortezomib
Drug: Doxorubicin
Drug: Dexamethasone

SUMMARY:
RATIONALE: Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as doxorubicin and dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) together with bortezomib may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving bortezomib together with doxorubicin and dexamethasone works in treating patients with multiple myeloma that has relapsed or not responded to treatment.

PATIENT POPULATION: Patients with relapsed or refractory multiple myeloma requiring therapy will be invited to participate in this study. Eligible patients will be >18 years old and able to give fully informed consent. Patients must have a Performance Score (PS) of 0-3 (ECOG), measurable serum and/or urine paraprotein, or serum free light chain, bilirubin value of less than one and a half times the upper limit of normal with ALT/AST values less than two and a half times the upper limit of normal. Patients with non-secretory multiple myeloma are excluded from this study.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the response (partial and complete response) in patients with relapsed or refractory multiple myeloma receiving bortezomib, doxorubicin hydrochloride, and dexamethasone (PAD) after prior treatment with a maximum of 6 courses of vincristine, doxorubicin, and dexamethasone (VAD) or VAD-like regimen.

Secondary

* To assess the safety and toxicity of PAD therapy in these patients.
* To determine the progression-free survival and overall survival of these patients.
* To compare the original response to VAD with the response obtained with PAD as assessed by percent fall in paraprotein or Bence Jones Protein, lowest level of abnormal protein achieved, and duration of response in these patients.

OUTLINE: This is a multicenter study.

STUDY DESIGN & METHODOLOGY:

This is a non-randomised, open labelled phase II trial in patients with relapsed or refractory multiple myeloma. Patients will be treated with: Bortezomib 1.3mg/m^2 bolus IV injection days 1, 4, 8 & 11 + Dexamethasone 40mg po on days 1, 2, 3, 4 + Doxorubicin 9mg/m^2/day IV continuous infusion over days 1 - 4. In addition, for the first cycle only, Dexamethasone will also be given at 40mg po on days 8 - 11 and 15 - 18.

Each treatment regimen will continue for a minimum of four - and up to six - cycles of 21 days (maximum response and 1 cycle).

This study planned to recruit a total of 69 patients in up to 8 centres in Ireland and the UK.

Patients will be enrolled in three groups of 23 patients:

* Relapsed patients, previously treated with VAD or VAD like regimen (VAMP, C-VAMP and Z-Dex are examples of VAD like therapy) and who have had autologous transplants at least 1 year previously. Patients may proceed directly to PAD therapy or have had a maximum of one other line of therapy before PAD.
* Relapsed patients, previously treated with VAD or VAD-like regimen who have not had autologous transplantation and achieved at least PR (Appendix A). Patients may proceed directly to PAD therapy or have had a maximum of two other lines of therapy before PAD.
* Patients refractory (MR, NC or PD) to VAD or VAD-like therapy. Patients should proceed directly to PAD therapy. Patients with NC or PD may proceed to PAD after a minimum of two cycles of VAD or VAD-like therapy or a minimum of 4 cycles, if MR.

After completion of study treatment, patients are followed every 2 months for 1 year.

ELIGIBILITY:
Inclusion criteria:

Each patient must meet all of the following inclusion criteria to be enrolled in the study:

1. Patients aged at least 18 years with MM requiring therapy for relapsed or refractory disease.
2. Previous VAD or VAD-like therapy (maximum 6 courses standard VAD). Subgroup allocation is shown in 4.1
3. Measurable serum and/or urine paraprotein, or serum free light chain
4. Performance Status (PS) 0-3 (ECOG - see Appendix B)
5. Serum bilirubin values <1.5 times the upper limit of normal
6. Serum ALT/AST values <2.5 times the upper limit of normal
7. Able to give informed consent

Exclusion criteria:

Patients meeting any of the following exclusion criteria are not to be enrolled in the study:

1. Females of child-bearing potential without a negative pregnancy test, immediately prior to the start of PAD therapy and/or unwilling to use barrier contraceptive precautions throughout the study or who are pregnant or breast-feeding
2. Men with partners of child bearing potential unwilling to use a medically acceptable form of contraception
3. Patients with non-secretory MM and no measurable elevation of serum free light chain
4. Performance status 4 (ECOG)
5. Patient has a platelet count <75 x 10^9/L within 14 days before enrolment
6. Patient has an absolute neutrophil count <1.0 x 10^9/L within 14 days before enrolment
7. Patient has a serum creatinine > 400 micromol/l at the time of enrolment
8. Patient has Grade 2 or greater than Grade 2 peripheral neuropathy or neuropathic pain as defined by NCI Common Terminology Criteria for Adverse Events version 3.0 (CTCAE) within 14 days before enrolment
9. Cardiac ejection fraction <40% by echocardiography or MUGA scan
10. Known HIV seropositivity (obligatory testing is not necessary)
11. Known Hepatitis B or C (obligatory testing is not necessary)
12. Patients who have received more than one autologous transplant
13. Use of any investigational drug within 4 weeks prior to enrolment or any patients scheduled to receive any investigational drug during the course of the study
14. Previous Bortezomib therapy
15. Patients who have a medical or psychiatric condition which, in the opinion of the investigator, contraindicates the patient's participation in this study
16. Previous or concurrent malignancies at other sites, with the exception of appropriately treated localized epithelial skin or cervical cancer. Patients with remote histories (>5 years) of other cured tumours may be entered
17. Plasma exchange within 21 days of enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2005-12; Primary Completion 2009-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Response rate (complete and partial response) | Patients will be followed in this study for approximately 16 months after recruitment to cover the period of PAD therapy plus one year follow up. The minimum frequency of reviews will be every two months.

SECONDARY OUTCOMES:
Progression-free survival | Patients will be followed in this study for approximately 16 months after recruitment to cover the period of PAD therapy plus one year follow up. The minimum frequency of reviews will be every two months.
Overall survival | Patients will be followed in this study for approximately 16 months after recruitment to cover the period of PAD therapy plus one year follow up. The minimum frequency of reviews will be every two months.
Compare original response to vincristine, doxorubicin, and dexamethasone with response to bortezomib, doxorubicin hydrochloride, and dexamethasone | Patients will be followed in this study for approximately 16 months after recruitment to cover the period of PAD therapy plus one year follow up. The minimum frequency of reviews will be every two months.

CONTACTS AND LOCATIONS:
Overall Officials: Curly Morris, Principal Investigator — Belfast City Hospital Trust Incorporating Belvoir Park Hospital
Locations (9):
- Ireland (5):
  - Adelaide and Meath Hospital, Dublin Incorporating the National Children's Hospital, Dublin
  - Mater Misericordiae University Hospital, Dublin
  - St. James's Hospital, Dublin
  - University College Hospital, Galway
  - Mid-Western Cancer Centre at Mid-Western Regional Hospital, Limerick
- United Kingdom (4):
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Saint Bartholomew's Hospital, London, England
  - University College Hospital, London, England
  - Belfast City Hospital Trust Incorporating Belvoir Park Hospital, Belfast, Northern Ireland